CLINICAL TRIAL: NCT04343976
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Pegylated Interferon Lambda vs. Placebo in Subjects Infected With COVID-19
Brief Title: Pegylated Interferon Lambda Treatment for COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to meet enrollment goal, lack of funding.
Sponsor: Raymond Chung (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Raymond Chung, Director of Hepatology, MGH, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P001083
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; COVID
Keywords: COVID; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lambda Treatment (Experimental): Treatment with subcutaneous injection (180 mcg) of pegylated interferon lambda
  Interventions: Drug: Pegylated interferon lambda
- Saline Placebo (Placebo Comparator): Subcutaneous injection of saline placebo
  Interventions: Drug: Pegylated interferon lambda

INTERVENTIONS:
Drug: Pegylated interferon lambda — 180 mcg subcutaneous injection of pegylated interferon lambda
  Other Names: Lambda

SUMMARY:
Prospective randomized trial to assess the antiviral efficacy of Pegylated Interferon Lambda (180 mcg SC injection) vs.placebo in up to 20 subjects with COVID-19 infection.

DETAILED DESCRIPTION:
The study objective is to assess the efficacy of Pegylated Interferon Lambda (180 mcg) vs. placebo in inducting quantitative PCR negativity at day 7

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Confirmed COVID-19 diagnosis based on PCR analysis of respiratory secretions
* Positive SARS-CoV-2 RT-PCR test must be within 48 hours of randomization

Exclusion Criteria:

* Clinically-significant illness or any other major medical disorder that in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol
* Treatment with IFN or other immunomodulatory/immunosuppressive agent within 12 months before screening.
* Respiratory compromise requiring ventilatory support other than nasal cannula (mask, bipap or intubation and mechanical ventilation)
* History of treatment with any of the following medications within five half-lives or 30 days before administration of the study drug (whichever is longer): anti-IL-6, anti-IL6R antagonists, Janus kinase inhibitors, ustekinumab (anti-IL-12/23), or anti IL-23 agents (guselkumab).
* Life threatening SAE during the screening period
* Pregnant or Nursing Females
* Platelet count <90,000 cells/mm3
* WBC count <3,000 cells/mm3
* ANC <1,500 cells/mm3
* Hb <11 g/dL for women and <12 g/dL for men
* CrCl < 50 mL/min
* Bilirubin level ≥ 1.5x ULN
* INR ≥1.5 (except in the setting of concomitant anticoagulant use)
* CRP > 200 mg/L
* Clinically-relevant alcohol or drug abuse within 12 months of screening
* Known hypersensitivity to Interferons
* Current or planned participation in an investigational new drug (IND) trial from 30-days prior to randomization through Day 14 post treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data is anticipated to be shared with outside institutions. Safety data will be shared with the drug manufacturer
Supporting Information: Study Protocol, ICF
Time Frame: Data is anticiapted to be made available within 3 months of study completion. Safety data, specifically treatment related adverse events, will be shared in real time
Access Criteria: researchers accessing IPD must be an approved and have a data use agreement in place with Partners Healthcare to access the data

REFERENCES:
- [Derived] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from inpatient admissions between June 2020 and July 2021.
Period: Overall Study
Arm/Group | Lambda Treatment | Saline Placebo
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lambda Treatment | Saline Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 54 [42 to 62] | 59 [40 to 72] | 54.5 [40 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Undetectable COVID PCR at Day 7
Description: Negative COVID PCR testing 7 days after first lambda dose
Time Frame: 7 days
Population: Subjects with Day 7 qPCR result of NEG (negative), meaning that no amplification was observed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lambda Treatment | Saline Placebo
Number analyzed (Participants) | 7 | 7
Participants | 1 | 4

2. Secondary Outcome: Undetectable COVID PCR at Day 3
Description: Negative COVID PCR testing 3 days after first lambda dose
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lambda Treatment | Saline Placebo
Number analyzed (Participants) | 7 | 6
Participants | 1 | 4

3. Secondary Outcome: Percentage of Subjects on Lambda vs Placebo With Symptomatic Improvement
Description: Daily symptom score improvement during treatment period
Time Frame: 2 weeks
Population: insufficient data, analysis not performed as there the symptom improvement score was not collected and not available for analysis.
Arm/Group | Lambda Treatment | Saline Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Subjects on Lambda vs Placebo With Improved Clinical Outcomes
Description: Time to event for death, intubation, hospital discharge
Time Frame: 2 weeks
Population: Data was not collected and therefor analysis not performed.
Arm/Group | Lambda Treatment | Saline Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Undetectable COVID PCR Testing at Day 14
Description: Negative COVID PCR testing 14 days after first lambda dose
Time Frame: 14 days
Population: All subjects providing NP swab samples at Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Lambda Treatment | Saline Placebo
Number analyzed (Participants) | 6 | 6
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collect beginning at time of consent (day 0) through study completion (day 14). Total period of 2 weeks.
Arm/Group | Lambda Treatment | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lambda Treatment (N=7) | Saline Placebo (N=7)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 4 lab abnormality
Worsening Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — required intubation prolonging hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lambda Treatment (N=7) | Saline Placebo (N=7)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 2
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — Grade 2
Stomach Pain (unspecified) (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3
ICU Delirium (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 2

LIMITATIONS AND CAVEATS:
Enrollment was slower than anticipated due to issues operationalizing outpatient follow-up for viremic subjects discharged from hospital prior to study completion, including lack of transportation and delays contracting with home health services to offer home visits. Also, study was terminated prior to meeting enrollment goal due to a decrease in eligible subjects and lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT04343976/Prot_SAP_000.pdf